CLINICAL TRIAL: NCT06195891
Title: A Single Center, Non-Randomized, Phase 1b Study of Orca-T Following Escalated Dose of Total Marrow and Lymphoid Irradiation in Patients With Acute Leukemias and MDS
Brief Title: Orca-T Following Chemotherapy and Total Marrow and Lymphoid Irradiation for the Treatment of Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia or Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23343; NCI-2023-08816 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23343 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-12-05; First posted 2024-01-08 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Specimen Handling; Biopsy; fludarabine; Magnetic Resonance Spectroscopy; Melphalan; Tacrolimus; Thiotepa; Lymphatic Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (TMLI, fludarabine, melphalan, Orca-T) (Experimental): PREPARATIVE REGIMEN: Patients undergo TMLI BID on days -8 to -5, followed by fludarabine IV on days -4 to -2 and melphalan IV on day -2. Patients receiving the lowest dose of TMLI also receive thiotepa IV on days -4 and -3.
  HCT: Patients receive Orca-T CD34+HSPC and Treg products IV on day 0, followed by the Orca-T tcon product IV on day 2.
  GVHD PROPHYLAXIS: Patients undergoing haplo-HCT receive tacrolimus starting on day 14 and continuing until day 90 with a taper per treating physician's discretion.
  Patients also undergo ECHO or MUGA scans, DECT/MRI scans, bone marrow biopsies/aspirates, and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Dual-Energy Computed Tomography; Procedure: Echocardiography; Drug: Fludarabine; Procedure: Magnetic Resonance Imaging; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Biological: Partially Engineered T-regulatory Cell Donor Graft TRGFT-201; Drug: Tacrolimus; Drug: Thiotepa; Radiation: Total Marrow and Lymphoid Irradiation

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Dual-Energy Computed Tomography — Undergo DECT/MRI scan
  Other Names: DECT
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Magnetic Resonance Imaging — Undergo DECT/MRI scan
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Partially Engineered T-regulatory Cell Donor Graft TRGFT-201 — Given IV
  Other Names: Orca-T; Partially Engineered and Enriched Treg Donor Graft TRGFT-201; T-cell-Depleted Graft With Additional Infusion of Conventional T Cells and Regulatory T Cells; TregGraft; TRGFT 201; TRGFT-201; TRGFT201
Drug: Tacrolimus — Given tacrolimus
  Other Names: FK 506; FK-506; Fujimycin; Hecoria; Prograf; Protopic; Tacforius
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Radiation: Total Marrow and Lymphoid Irradiation — Undergo TMLI
  Other Names: TMLI

SUMMARY:
This phase I trial tests the side effects and best dose of total marrow lymphoid irradiation along with chemotherapy, with fludarabine and melphalan, with or without thiotepa, in combination with Orca-T cells for patients with acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL) or myelodysplastic syndrome (MDS). Total marrow and lymphoid irradiation is a targeted form of total body irradiation that uses intensity-modulated radiation therapy to target marrow, lymph node chains, and the spleen. It is designed to reduce radiation-associated side effects and maximize the radiation therapeutic effect. Giving chemotherapy with medications such as thiotepa, fludarabine, and melphalan before a treatment with stem cells helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. Orca-T cells take cells from a donor and remove some of the T cells and replace them with partially engineered T cells in order to induce better tolerance in patients. Giving total marrow and lymphoid irradiation and chemotherapy followed by Orca -T cells may be an effective treatment for patients with AML, ALL or MDS.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Describe toxicities attributable to total marrow and lymphoid irradiation (TMLI) by dose level in patients with high-risk acute leukemias or MDS, in the context of partially engineered T-regulatory cell donor graft TRGFT-201 (Orca-T) from a matched or haploidentical donor.

II. Determine the recommended phase II dose (RP2D) of TMLI with an Orca-T for allogeneic hematopoietic cell transplantation (HCT).

SECONDARY OBJECTIVES:

I. Determine incidence of acute and late HCT-related immune complications (infections, etc.) at 100 days and 1 year.

II. To evaluate the safety of the regimen, at each dose level, by assessing the following: type, frequency, severity, attribution, time course and duration of adverse events in dose limiting toxicity (DLT) window of 28 days at each dose level, including acute graft-versus-host disease (GVHD), infection and delayed engraftment within the first 100 days and chronic GVHD incidence at 1 year.

III. Measure incidence of acute and chronic GVHD at 100 days and 1-year post-HCT, respectively.

IV. Measure GVHD-free and relapse-free survival (GRFS) at 1-year post-HCT.

EXPLORATORY OBJECTIVES:

I. Estimate overall survival (OS), event-free survival (EFS), cumulative incidence (CI) of relapse/progression, and non-relapse mortality (NRM) at 100 days, 1 year and 2 years.

II. Evaluate the effect of TMLI as conditioning for Orca-T HCT on immune reconstitution at 1, 3, 6, 9 and 12 months after alloHCT.

III. Evaluate GVHD biomarkers and inflammatory cytokines on days +7, +14, and +30, (all patients) and upon GVHD onset/resolution.

IV. Investigate the temporal effect and bone marrow residual damage and regeneration on days +30, +100, and 1-year post-alloHCT by using longitudinally collected biological samples and imaging.

V. Monitor effects of TMLI as conditioning on gastrointestinal (GI) toxicity and T cell signaling pathways.

VI. Monitor effects of TMLI on GI microbiome diversity.

OUTLINE: This is a dose-escalation study of TMLI followed by a dose-expansion study.

PREPARATIVE REGIMEN: Patients undergo TMLI twice a day (BID) on days -8 to -5, followed by fludarabine intravenously (IV) on days -4 to -2 and melphalan IV on day -2. Patients receiving the lowest dose of TMLI also receive thiotepa IV on days -4 and -3.

HCT: Patients receive Orca-T CD34+hematopoietic stem and progenitor cells (HSPC) and T-regulatory cell (Treg) products IV on day 0, followed by the Orca-T conventional t-cell (tcon) product IV on day 2.

GVHD PROPHYLAXIS: Patients undergoing haploidentical (haplo)-HCT receive tacrolimus starting on day 14 and continuing until day 90 with a taper per treating physician's discretion.

Patients also undergo echocardiogram (ECHO) or multigated acquisition (MUGA) scans, dual energy computed tomography (DECT)/magnetic resonance imaging (MRI) scans, bone marrow biopsies/aspirates, and blood sample collection throughout the study.

After completion of study treatment, patients are followed for up to 2 years from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant
* Agreement to allow the use of archival tissue from diagnostic bone marrow biopsies

  * If unavailable, exceptions may be granted with study primary investigator (PI) approval
* Age: 60-75 years
* Karnofsky performance status ≥ 70
* Eligible patients will have a histopathological confirmed diagnosis of hematologic malignancy in one of the following categories:

  * Acute myelogenous leukemia:

    * Patients with de novo or secondary disease in CR1 or more with European LeukemiaNet (ELN) intermediate or adverse risk category, or
    * Patients with active disease

      * Morphologically; or
      * Minimal residual disease (MRD) + (flow cytometry of ≥ 0.1%, next generation sequencing [NGS] or cytogenetics)
  * Acute lymphoblastic leukemia (ALL):

    * Patients with de novo or secondary disease according to National Comprehensive Cancer Network (NCCN) guidelines for ALL hypoploidy (< 44 chromosomes); t(v;11q23): MLL rearranged; t(9;22) (q34;q11.2); complex cytogenetics (5 or more chromosomal abnormalities); high white blood cell (WBC) at diagnosis (≥ 30,000 for B lineage or ≥ 50,000 for T lineage); iAMP21loss of 13q, and abnormal 17p; or
    * Patients with active disease:

      * Morphologically; or
      * MRD+ (flow cytometry of ≥ 0.1%, or cytogenetics)
  * Myelodysplastic syndrome in high-intermediate (int-2) and high risk categories per International Prognostic Scoring System Risk (IPSSR)
* Serum direct (conjugated) bilirubin ≤ 2.0 mg/dl performed within 30 days prior to day 1
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 times the institutional upper limits of normal performed within 30 days prior to day 1. Patients with Gilberts disease are allowed
* Creatinine clearance of ≥ 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula performed within 30 days prior to day 1
* Ejection fraction measured by echocardiogram or MUGA ≥ 50% performed within 30 days prior to day 1
* If able to perform pulmonary function tests: forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and carbon monoxide diffusing capability (DLCO) (diffusion capacity) ≥ 50% of predicted (corrected for hemoglobin).

If unable to perform pulmonary function tests: oxygen (O2) saturation > 92% on room air performed within 30 days prior to day 1

* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test performed within 30 days prior to day 1. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* PATIENTS: Patients should have discontinued all previous intensive therapy, chemotherapy or radiotherapy for 2 weeks prior to commencing therapy on this study NOTE: Low dose chemotherapy or maintenance chemotherapy given within 7 days of planned study enrollment is permitted. These include hydroxyurea, 6-meraptopurine, oral methotrexate, vincristine, oral etoposide, and tyrosine kinase inhibitors (TKIs). FLT-3 inhibitors can also be given up to 3 days before conditioning regimen.) All patients with prior radiation treatment to the lung, liver, and kidney will be excluded. For other scenarios of prior radiation treatment, up to 2000 cGy at 2 Gy per day will be allowed. Inclusion of patients with previous radiation exposure will be determined based on the radiation oncologist medical doctor (MD) evaluation and judgment
* DONORS: All candidates for this study must have an human leukocyte antigen (HLA) (A, B, C, and DR) identical sibling who is willing to donate mobilized peripheral blood stem cells or have a 10/10 (A, B, C, DR and DQ) allele matched unrelated donor (DQ or DP mismatch is allowed per discretion of the principal investigator), or haploidentical donor. City of Hope (COH) standard operating procedures (SOP) (B.001.11) will be used for allogeneic donor evaluation, selection, and consent. Donor screening will be in compliance with all requirements of Food and Drug Administration (FDA) regulation 21 Code of Federal Regulations (CFR) Part 1271 including donor screening for COVID-19 exposure or infection

Exclusion Criteria:

* PATIENTS: Prior allogeneic stem cell transplant
* PATIENTS: More than 3 prior lines of intensive chemotherapy, where the regimen intent was to induce remission
* PATIENTS: Receiving any other investigational agents or concurrent biological, intensive chemotherapy or radiation therapy for the previous 2 weeks from conditioning NOTE: Low dose chemotherapy or maintenance chemotherapy given within 7 days of planned study enrollment is permitted. These include: Hydroxyurea, 6-meraptopurine, oral methotrexate, vincristine, oral etoposide, and tyrosine kinase inhibitors (TKIs). FLT-3 inhibitors can also be given up to 3 days before conditioning regimen
* PATIENTS: History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* PATIENTS: Having any uncontrolled illness including ongoing or active bacterial, viral or fungal infection requiring antibiotics
* PATIENTS: Patients with other active malignancies are ineligible for this study, other than non-melanoma skin cancer, in situ cervical cancer and prostate cancer. Patients with prior history of localized prostate cancer treated with curative intent regardless of time from the treatment to study entry, and patients with prostate cancer receiving active surveillance not requiring therapy are eligible
* PATIENTS: The recipient has a medical problem or neurologic/psychiatric dysfunction which would impair his/her ability to be compliant with the medical regimen and to tolerate transplantation or would prolong hematologic recovery which in the opinion of the principal investigator would place the recipient at unacceptable risk
* PATIENTS: Females only: Pregnant or breastfeeding
* PATIENTS: Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* PATIENTS: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2027-06-21 (Estimated); Study Completion 2027-06-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From start of conditioning to day +100
  Will be scored on both the Bearman Scale and National Cancer institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5 scale.

SECONDARY OUTCOMES:
Relapse/progression rate | From start of therapy to relapse/progression, up to 2 years
  The event is relapse/progression. Time to this event is measured from start of therapy. Death without relapse/progression is considered a competing risk. Surviving patients with no history of relapse/progression are censored at time of last follow-up.
Non-relapse mortality | From start of therapy until non-disease related death, disease relapse/progression, whichever comes first, up to 2 years
  Will be calculated using the Kaplan-Meier method.
Incidence of infection | From day 0 to day +100
  Will be reported by site of disease, date of onset, severity and resolution, if any.
Incidence of adverse events | From day -9 to day +100
  Toxicities of grade 3, 4, or 5 per Bearman Scale and CTCAE v5.0.
Acute graft versus host disease (GVHD) of grades 2-4 and 3-4 | From date of stem cell infusion to document/biopsy proven acute GVHD onset date (within the first 100 days post-transplant)
  Documented/biopsy proven acute graft versus host disease is graded according to the 2016 consensus grading.
Chronic Graft versus Host Disease rate | From approximately 80-100 days post-transplant to the documented/biopsy proven chronic GVHD, up to 2 years
  Documented/biopsy proven chronic graft versus host disease (cGvHD) is scored. Time to event is measured from approximately 80-100 days post-transplant to the documented/biopsy proven chronic GVHD onset date and will be used to estimate the cumulative incidence. Relapse/NRM will be competing risk events for cGVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Salhotra, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States